CLINICAL TRIAL: NCT06648317
Title: Radiolabelled Nectin-4 Targeted LMW Probe PET/CT in Patients With Lung Lesions
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, nanli, Professor, Peking University Cancer Hospital & Institute
Other Study IDs: 2022KT37-ZY01-1
Record Dates: First submitted 2024-09-24; First posted 2024-10-18 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer, Non-Small Cell; Lung Infection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FDG-PET — All study participants will undergo 18F-FDG PET/CT scan within 1 week

SUMMARY:
To evaluate the ability of [68Ga]N188 to detect nectin-4 overexpression in patients with lung lesions.

DETAILED DESCRIPTION:
To evaluate the ability of [68Ga]N188 to detect nectin-4 overexpression in patients with different lung lesions, such as inflammation and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female;
2. Heart function is normal;
3. Normal heart function;
4. Estimated survival ≥12 weeks;
5. Good follow-up compliance;
6. presence of at least one measurable target lesion according to RECIST1.1 criteria;
7. Women of childbearing age (15-49 years) must have a negative pregnancy test within 7 days before starting the test; Fertile men and women must agree to use effective contraception to prevent pregnancy during the study period and for 3 months after the test;
8. Patients recommended by clinicians to undergo PET/CT examination for tumor diagnostic staging;
9. The subject patients could fully understand and voluntarily participate in the experiment, and signed the informed consent.

Exclusion Criteria:

1. Serious abnormality of liver, kidney and blood;
2. Pregnant patients;
3. Pregnant and lactation women;

3) unable to lie flat for half an hour; 4) Refuse to join the clinical investigator; 5) Suffering from claustrophobia or other mental diseases; 6) Other conditions that researchers deem unsuitable for participating in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lung lesions
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 1 year
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions. The uptake of the tracer （68Ga-N188） in lung lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Li, MD, Principal Investigator — Peking University Cnacer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No